CLINICAL TRIAL: NCT01014351
Title: A Phase II Study of Everolimus in Combination With Paclitaxel and Carboplatin in Patients With Metastatic Melanoma
Brief Title: Study of Everolimus With Paclitaxel and Carboplatin in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI MEL 19
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-01

CONDITIONS: Metastatic Melanoma
Keywords: Metastatic Melanoma; Everolimus; Paclitaxel; Carboplatin
MeSH Terms: conditions — Melanoma | interventions — Paclitaxel; Carboplatin; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel/Carboplatin/Everolimus (Experimental): Systemic Therapy using everolimus, paclitaxel and carboplatin given during a 21-day treatment cycle
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Everolimus

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel, 175mg/m2 by IV infusion over 1-3 hours on day 1 of every 21 day cycle
  Other Names: Taxol
Drug: Carboplatin — Carboplatin, AUC 6 given by IV infusion over 20-30 minutes on day 1 of every 21 day cycle
  Other Names: Paraplatin
Drug: Everolimus — Everolimus, 5 mg by mouth (PO) once a day, continuous dosing every 21-day cycle
  Other Names: RAD001; Afinitor

SUMMARY:
Based on data demonstrating synergy between paclitaxel and mammalian target of rapamycin (mTOR) inhibition, the investigators propose that the addition of everolimus to paclitaxel with carboplatin should lead to improvements in efficacy as measured by progression-free survival and response rate.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic melanoma.
2. Stage III or IV disease that is not amenable to resection.
3. Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. If the patient has had previous radiation to the target lesion(s), there must be evidence of progression since the radiation.
4. ECOG Performance Status of 0 or 1.
5. Life expectancy ≥12 weeks.
6. No prior cytotoxic chemotherapy or targeted therapy. Immunotherapy is allowed (i.e., interleukin-2 or interferon).
7. Adequate hematological function:

   * absolute neutrophil count (ANC) ≥1500/µL and
   * platelets ≥100,000/µL and
   * hemoglobin >9 g/dL
8. Adequate renal function: serum creatinine ≤2.0 mg/dL or calculated (measured) GFR ≥50 mL/min.
9. Adequate hepatic function:

   * serum bilirubin ≤1.5 x institutional upper limit of normal (ULN);
   * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN, or ≤5 × ULN in patients with documented liver metastases.
10. Normal PT, INR. Patients on coumadin anticoagulation are eligible if they are on a stable dose, with an INR in the therapeutic range.
11. Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can be included after initiation of appropriate lipid lowering medication.
12. Age ≥18 years.
13. Ability to swallow whole pills.
14. Patient must be accessible for treatment and follow-up.
15. Patients must be able to understand the investigational nature of this study and give written informed consent prior to study entry.

Exclusion Criteria:

1. Previous treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus), paclitaxel, or carboplatin.
2. Treatment with any investigational agent ≤4 weeks of protocol treatment.
3. Patients currently receiving anticancer therapies or who have received anticancer therapies ≤3 weeks of the start of the study drug (including radiation therapy, immunotherapy).
4. Patients, who have had a major surgery or significant traumatic injury ≤4 weeks of start of study drug or patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia).
5. Patients receiving chronic, systemic treatment with corticosteroids (dose >10 mg daily of methylprednisolone or equivalent) or other immunosuppressive agents. Topical or inhaled steroids are allowed.
6. Immunization with attenuated live vaccine ≤1 week of study or anytime during study treatment period.
7. Patients with active brain metastases are ineligible. Patients with treated brain metastases are eligible if (1) radiation therapy was completed ≥4 weeks prior to study entry; (2) surgery was completed ≥4 weeks prior to study entry; (3) follow-up scan shows no disease progression; and (4) patient does not require steroids.
8. Any severe and/or uncontrolled medical conditions or other conditions that could affect participation in the study such as:

   * severely impaired lung function defined as a DLCO ≤50% of the normal predicted value and/or O2 saturation ≤88% at rest on room air.
   * symptomatic congestive heart failure of New York Heart Association Class III or IV.
   * unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant disease.
   * uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN.
   * active (acute or chronic) uncontrolled severe infections.
   * liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis.
9. Active, bleeding diathesis.
10. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
11. A known history of human immunodeficiency virus (HIV) seropositivity.
12. Known hypersensitivity to everolimus or other rapamycins (sirolimus, temsirolimus) or to its excipients.
13. Use of St. John's Wort is prohibited. Drugs or substances (e.g., grapefruits, star fruits, seville oranges, and their juices and products), known to be inhibitors or inducers of the isoenzyme CYP3A4 should be avoided. Co-administration with substrates, inducers, or inhibitors of P glycoprotein should also be avoided.
14. Female patients who are pregnant or breastfeeding or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes. Hormonal contraceptives are not acceptable as a sole method of contraception. (Women of childbearing potential [WOCBP] must have a negative urine or serum pregnancy test within 7 days prior to administration of everolimus.) WOCBP should continue to use effective contraception for 8 weeks after ending everolimus treatment.
15. Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
16. History of noncompliance to medical regimens. Patients unwilling to, or unable to, comply with the protocol.
17. History of any other disease, physical examination finding, or clinical laboratory finding that gives reasonable suspicion of a disease or a condition that may render the patient at high risk for treatment complications using these agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (12):
- United States (12):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Oncology Hematology of SW Indiana, Evansville, Indiana
  - Hematology Oncology Clinic, LLP, Baton Rouge, Louisiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Grand Rapids Oncology Program, Grand Rapids, Michigan
  - Research Medical Center, Kansas City, Missouri
  - Nebraska Methodist Cancer Center, Omaha, Nebraska
  - Oncology Hematology Care, Cincinnati, Ohio
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Peninsula Cancer Institute, Newport News, Virginia

REFERENCES:
- [Result] Hauke RJ, Infante JR, Rubin MS, Shih KC, Arrowsmith ER, Hainsworth JD. Everolimus in combination with paclitaxel and carboplatin in patients with metastatic melanoma: a phase II trial of the Sarah Cannon Research Institute Oncology Research Consortium. Melanoma Res. 2013 Dec;23(6):468-73. doi: 10.1097/CMR.0000000000000014. PMID 23969699
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=23969699

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paclitaxel/Carboplatin/Everolimus
Started | 70
Completed | 33
Not Completed | 37

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel/Carboplatin/Everolimus
Number analyzed (Participants) | 70
Age, Continuous [Median (Full Range); unit: years] | 63 [29 to 82]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 46
Region of Enrollment [Number; unit: participants]
  United States | 70

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time from randomization until objective tumor progression (PD) or death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Paclitaxel/Carboplatin/Everolimus
Number analyzed (Participants) | 70
Months | 4.04 [2.76 to 4.99]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from randomization until death from any cause.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Paclitaxel/Carboplatin/Everolimus
Number analyzed (Participants) | 70
Months | 10.12 [7.29 to 10.87]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) is defined as the Percentage of Patients Who Experience an Objective Benefit From Treatment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 18 months
Measure: Number; unit: percentage of patients
Arm/Group | Paclitaxel/Carboplatin/Everolimus
Number analyzed (Participants) | 70
percentage of patients | 17

ADVERSE EVENTS:
Arm/Group | Paclitaxel/Carboplatin/Everolimus
Serious Adverse Events (participants affected / at risk) | 29/70
Other Adverse Events (participants affected / at risk) | 70/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel/Carboplatin/Everolimus (N=70)
Acute angioedema (Vascular disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4)
Fever (General disorders) | 3 (3)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 3 (3)
Hemorrhage, CNS (Nervous system disorders) | 1 (1)
Hemorrhage, GI (Gastrointestinal disorders) | 2 (2)
Hemorrhage, pulmonary/upper respiratory - nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Infection - bone (osteomyelitis) (Infections and infestations) | 1 (2)
Infection - lung (pneumonia) (Infections and infestations) | 1 (1)
Mental status (Psychiatric disorders) | 1 (1)
Muscle weakness - extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness - generalized (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Thrombosis/embolism (vascular access) (Vascular disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 6 (7)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel/Carboplatin/Everolimus (N=70)
Fatigue (General disorders) | 53
Hemoglobin (Blood and lymphatic system disorders) | 46
Platelets (Investigations) | 39
Nausea (Gastrointestinal disorders) | 38
Neutrophils/granulocytes (Investigations) | 33
Hair loss/alopecia (Skin and subcutaneous tissue disorders) | 32
Neuropathy: sensory (Nervous system disorders) | 31
Leukocytes (total WBC) (Investigations) | 30
Rash/desquamation (Skin and subcutaneous tissue disorders) | 27
Diarrhea (Gastrointestinal disorders) | 27
Constipation (Gastrointestinal disorders) | 24
Triglyceride, serum-high (Metabolism and nutrition disorders) | 22
Anorexia (Metabolism and nutrition disorders) | 21
Mucositis/stomatitis (Gastrointestinal disorders) | 21
Vomiting (Gastrointestinal disorders) | 20
Glucose, serum-high (Metabolism and nutrition disorders) | 20
Muscle weakness (Musculoskeletal and connective tissue disorders) | 19
Cholesterol, serum-high (Investigations) | 17
Pain - bone (Musculoskeletal and connective tissue disorders) | 16
Pain - joint (Musculoskeletal and connective tissue disorders) | 15
Edema (General disorders) | 15
Pain - muscle (Musculoskeletal and connective tissue disorders) | 14
Weight loss (Investigations) | 13
Dizziness (Nervous system disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Creatinine (Metabolism and nutrition disorders) | 12
Fever (General disorders) | 12
Taste alteration (dysgeusia) (Nervous system disorders) | 11
Insomnia (Psychiatric disorders) | 11
Pain (General disorders) | 10
Hemorrhage, pulmonary/upper respiratory - nose (Respiratory, thoracic and mediastinal disorders) | 10
Alkaline phosphatase (Investigations) | 10
Calcium - serum-low (Metabolism and nutrition disorders) | 10
Paresthesia (Nervous system disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Thrombosis/thrombus/embolism (Vascular disorders) | 9
Dehydration (Metabolism and nutrition disorders) | 9
Sodium, serum-low (Metabolism and nutrition disorders) | 9
Pruritus/itching (Skin and subcutaneous tissue disorders) | 8
Pain - abdomen NOS (Gastrointestinal disorders) | 8
Rigors/chills (General disorders) | 7
Pain - extremity (Musculoskeletal and connective tissue disorders) | 7
Dermatology/skin - other (Skin and subcutaneous tissue disorders) | 7
Pain - head (Nervous system disorders) | 7
AST, SGOT (Investigations) | 7
ALT, SGPT (Investigations) | 6
Potassium, serum-low (Metabolism and nutrition disorders) | 6
Infection (Infections and infestations) | 6
Mood alteration - depression (Psychiatric disorders) | 6
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 5
Mood alteration - anxiety (Psychiatric disorders) | 5
Pain - back (Musculoskeletal and connective tissue disorders) | 5
Hyperlipidemia (Metabolism and nutrition disorders) | 5
Potassium, serum-high (Metabolism and nutrition disorders) | 5
Pain - throat (Respiratory, thoracic and mediastinal disorders) | 4
Ocular/visual - other (Eye disorders) | 4
Albumin, serum-low (Metabolism and nutrition disorders) | 4
Bicarbonate, serum-high (Metabolism and nutrition disorders) | 4
Magnesium, serum-low (Metabolism and nutrition disorders) | 4
Pain - chest (General disorders) | 4
BUN levels decreased (General disorders) | 4
Flushing (Vascular disorders) | 4
BUN levels increased (General disorders) | 4
Hypobilirubinemia (Investigations) | 4
Nasal drainage (Respiratory, thoracic and mediastinal disorders) | 4
Extremity-lower (gait/walking) (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.